CLINICAL TRIAL: NCT00391950
Title: An Open-Label, Randomized, Multicentre Study to Evaluate the Efficacy of Two Zoledronic Acid Schedules on Bone Mineral Density in Prostate Cancer Patients Undergoing Androgen Deprivation Therapy
Brief Title: Maintaining Bone Strength in Men With Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GGB12
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Cancer treatment induced bone loss (CTIBL); Androgen deprivation therapy (ADT)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
The purpose of this study is to see if giving zoledronic acid three times a year is as effective as five times a year, in increasing bone strength in men with prostate cancer. All participants will receive the active drug but half will receive drug every 6 months and the other half will receive drug every 3 months. Both patient and doctor will know which treatment a patient is receiving.

After 1 year of treatment bone strength will be measured with scans and compared to the strength at the start of the study. All participants will stop receiving the drug after 1 year and will be seen back in the clinic, annually for another 2 years for follow-up.

ELIGIBILITY:
Inclusion criteria:

Histologically confirmed diagnosis of carcinoma of the prostate

* No distant metastases
* Patients must be candidates for androgen deprivation therapy (ADT)
* Patient with a baseline BMD T-score at or below -1 standard deviations in the lumbar spine (L2-L4) are eligible

Exclusion criteria:

Patients with normal BMD at trial entry

* Patients who received any prior bisphosphonate therapy in the past 12 months
* Treatment with anti-androgen mono- or combination therapy
* Patients who are currently receiving diethylstilbesterol (DES) or who have previously received PC-SPES
* Patients who have received prior treatment with systemic corticosteroids within the past 12 months
* Patients with prior exposure to anabolic steroids or growth hormone within the past 6 months
* Patients with any prior treatment for osteoporosis

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density (BMD) at lumbar spine as assessed by dual energy x-ray absoptiometry (DEXA) scan

SECONDARY OUTCOMES:
To compare the effect of zoledronic acid 4 mg every 12 weeks versus every 24 weeks on:
The percent change in BMD of the total hip following one year of therapy and the forearm following one year of therapy. This will be carried out at a limited number of centres.
Quality of life following one year of therapy.
Various biochemical markers of bone resorption (N-telopeptide, NTX, C-telopeptide, CTX, TRACP, PINP) and bone formation (bone alkaline phosphatase, BAP) during one year of therapy. This will be carried out at a limited number of centres.
Percentage of and rate of vertebral and hip fractures.
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Derby, United Kingdom